CLINICAL TRIAL: NCT01729936
Title: Effectiveness of an Intervention to Reduce Diary Hours of Sitting Time in Overweight and Obese Patients (SEDESACTIV):Simple Randomized Controlled Trial
Brief Title: SedestActiv Project: Intervention to Reduce Diary Hours of Sitting Time in Overweight and Obese Patients
Acronym: SedestActiv
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fondo de Investigacion Sanitaria (Other); Preventive Services and Health Promotion Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI11/01082
Record Dates: First submitted 2012-08-01; First posted 2012-11-21 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Overweight; Obese; Sedentary
Keywords: Sitting time; Overweight; Obese; Primary Health Care
MeSH Terms: conditions — Overweight; Obesity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitting time Change Intervention (Experimental): Sitting time Change Intervention: recommendation to substitute Sitting time by doing the regular activities standing or walking.
  Duration: 6 month. Frequency: 1 time each 15 days during the first 4 month and 1 time each month the last 2 months.
  Interventions: Behavioral: Sitting time Change Intervention
- Active Control (No Intervention): Control visits to the Primary Health Care Center

INTERVENTIONS:
Behavioral: Sitting time Change Intervention — Intervention to find alternatives to substitute sitting time by doing the regular activities standing or walking.
  Other Names: SedestActiv Intervention
  Arms: Sitting time Change Intervention

SUMMARY:
Primary care centres are a key setting to treat people with overweight and moderate obesity. There is growing evidence that sitting for a long time is negatively associated with people's health. Interventions with the aim of reducing daily time of sedentary activities can be an effective strategy to increase daily energy expenditure. To improve the effectiveness of programmes promoting physical activity in primary care we need some clear action protocols that can be easily integrated in the daily routines of primary care professionals.

Objective. The objective of the study is to evaluate the effectiveness of a six-moth primary care intervention to reduce diary hours of sitting time in overweight and obese sedentary patients, as well as to increase their weekly caloric spend.

Methods. The design of the study is a simple randomized controlled trial. Ten primary care centers will be invited to participate and will be randomized into control (CG) and intervention group (IG). Each professional will randomly invite to participate voluntarily moderate obese or overweight patients (BMI: 25-34,9 kg/m2) of both sexes, aged between 25 and 65 years old, who are 6 or more than 6 hours daily sitting. A total of 400 subjects (200 individuals in each group) are needed. In addition, 50 subjects with fibromyalgia will be included in the study to know the feasibility of the intervention among them.

The main dependent variable (sitting times) will be measured with an ActivPAL during first and last intervention week. There will be a follow up after 3, 6 and 12 months of the end of the intervention. Other variables included in the study: number of steps walked, subjective level of physical activity, weight, height, BMI, skinfolds, waist circumference, triglycerides, total cholesterol, (LDL and HDL), glucose, sociodemographic variables, blood pressure and quality of life related to health. A descriptive analysis of all variables and a multivariate analysis to assess differences among intervention and control group will be undertaken. Multivariate analysis will be carried out to assess time changes of dependent variables. All the analysis will be done under the intention to treat principle.

DETAILED DESCRIPTION:
The intervention will be based on a recommendation to find alternatives to progressively substitute Sitting time by doing the regular activities standing or walking. Control group will receive minimum advice.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and moderate obese patients (BMI: 25-34,9 kg/m2).
* Be 6 or more than 6 hours daily sitting.
* Able to walk and stand up from a chair unaided.
* Subjects who can guarantee a year continuity in the study.

Exclusion Criteria:

* Recommended contradictions to advising physical activity to overweight and obese people.
* Have an obesity surgical operation.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-02 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of a 6-month primary care intervention to reduce diary hours of Sitting time in overweight and obese patients, as well as to increase their weekly caloric spend | Baseline-6-9-12 and 18 month
  In this part of the study will use two measure tools: 1) A sitting time test during a working day and during the weekends (Marshall Test). 2) The activPal device will measure the sitting, stand and walking minutes and Mets expended during a week period.

SECONDARY OUTCOMES:
Number of steps walked | Baseline-6-9-12 and 18 month
Subjective level of physical activity | Baseline-6-9-12 and 18 month
Quality of life related to health | Baseline-6-9-12 and 18 month
Blood pressure | Baseline-6-9-12 and 18 month

OTHER OUTCOMES:
Skinfolds and waist circumference | Baseline-6-9-12 and 18 month
Triglycerides, total cholesterol and glucose | Baseline-6-9-12 and 18 month

CONTACTS AND LOCATIONS:
Overall Officials: Martínez R Elena, Principal Investigator — Institut Català de la Salut
Locations (1):
- IDIAP Jordi Gol, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Rodriguez-Roca B, Urcola-Pardo F, Anguas-Gracia A, Subiron-Valera AB, Gasch-Gallen A, Anton-Solanas I, Gascon-Catalan AM. Impact of Reducing Sitting Time in Women with Fibromyalgia and Obesity: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jun 9;18(12):6237. doi: 10.3390/ijerph18126237. PMID 34207661
- [Derived] Martin-Borras C, Gine-Garriga M, Martinez E, Martin-Cantera C, Puigdomenech E, Sola M, Castillo E, Beltran AM, Puig-Ribera A, Trujillo JM, Pueyo O, Pueyo J, Rodriguez B, Serra-Paya N; SEDESTACTIV Study Group. Effectiveness of a primary care-based intervention to reduce sitting time in overweight and obese patients (SEDESTACTIV): a randomized controlled trial; rationale and study design. BMC Public Health. 2014 Mar 5;14:228. doi: 10.1186/1471-2458-14-228. PMID 24597534